CLINICAL TRIAL: NCT05808738
Title: The Effect of Therapeutic Gaming Used in Preparation for Hydrothera-py Treatment on Children's Pain, Fear and Emotional Indicators: A Ran-domized, Controlled, Treatment Study
Brief Title: The Effect of Therapeutic Play on Pain, Fear and Emotional Indicator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Elif Nilay Kizilay, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: DOKTORA TEZ
Record Dates: First submitted 2023-01-08; First posted 2023-04-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Hydrotherapy
Keywords: hyrotherapy; therapeutic game; child
MeSH Terms: interventions — Play Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic game group (Active Comparator): therapeutic play will be played 10 minutes before the hydrotherapy treatment.
  Interventions: Behavioral: therapeutic play
- control group (No Intervention): No intervention was given to the children prior to hydrotherapy treatment.

INTERVENTIONS:
Behavioral: therapeutic play — therapeutic game will be played to prepare children for hydrotherapy treatment
  Arms: therapeutic game group

SUMMARY:
This study was planned to determine the effect of therapeutic play and preparation for hydrotherapy treatment on pain, fear and emotional indicator levels in children with burn injuries.

It is an experimental randomized controlled study. The population of the research will be children between the ages of 3-6 who are hospitalized in the Pediatric Burn Intensive Care Unit. As a result of the power analysis using the G*Power 3.0.10 program, at least 52 children in total (control group 26, therapeutic play group 26) with 50% power, 0.05 alpha margin of error, 0.80 beta margin of error and 20% effect size. was determined to be included in the study. However, considering the case losses, the number of children to be included in the study was determined as 64 by increasing the sample size by 20%. The data will be collected between the dates to be determined by the researcher after obtaining the ethics committee approval and written permission from the institution where the research will be conducted. Introductory information form, FLACC Pain Scale, Child Fear Scale and Child Emotional Indicators Scale will be used to collect research data.

The research will be conducted with the children of parents who agreed to participate in the study. There are two groups, the control group and the experimental group. While the routine practice of the clinic will be applied to the control group, creative therapeutic games will be played to the experimental group together with the routine practice. Children will be stratified according to their pain scores, fear scores and burn depth (degree) and will be assigned to an equal number of children in each group using the blocking method. Before the procedure, the introductory information form will be filled in by the researcher in line with the patient file and parent information. After parents are informed about which group the child is in, their written consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 3-6 years old
* The child is receiving the first hydrotherapy treatment in the clinic.
* Presence of second and/or third degree superficial and/or deep burns
* Volunteering of the child and family to participate in the research
* The child was given analgesics half an hour before the procedure.
* No simultaneous debridement during hydrotherapy
* Burn width between 20%-70%

Exclusion Criteria:

* The child is younger than 3 years old, over 6 years old
* Presence of any other chronic disease other than burns
* The child is receiving mechanical ventilator support.
* Having a trecheostomy done to the child
* The child has been given sedative medication in the last 8 hours.
* Having a companion other than mother or father
* Hydrotherapy treatment takes less than 30 minutes, more than 45 minutes
* The child does not want to play

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The change in the pain level of the children will be evaluated by applying the FLACC pain scale to the children by the researcher. | Pain assessment will be done 30 minutes before hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment
The change in the pain level of the children will be evaluated by applying the FLACC pain scale to the children by the researcher. | Pain assessment will be done 10 minutes after hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment
The change in the pain level of the children will be evaluated by applying the FLACC pain scale to the children by the researcher. | Pain assessment will be done 30 minutes after hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment

SECONDARY OUTCOMES:
The change in the children's fear level will be evaluated by applying the Child Fear Scale to the children by the researcher. | Fear assessment will be done 30 minutes before hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment
The change in the children's fear level will be evaluated by applying the Child Fear Scale to the children by the researcher. | Fear assessment will be done 10 minutes after hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment
The change in the children's fear level will be evaluated by applying the Child Fear Scale to the children by the researcher. | Fear assessment will be done 30 minutes after hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment

OTHER OUTCOMES:
The change in children's emotional status will be evaluated by applying the Children's Emotional Indicators Scale to the children by the researcher. | Emotional indicators will be evaluated at the 10th minute of hydrotherapy treatment.
  therapeutic game was played for children 10 minutes before hydrotherapy treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No